CLINICAL TRIAL: NCT04205929
Title: Treatment of Unfavorable Bleeding Patterns in Contraceptive Implant Users: a Randomized Clinical Trial of Curcumin
Brief Title: Use of Curcumin to Treat Unfavorable Bleeding Patterns in Contraceptive Implant Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Alison Edelman, Professor OB/Gyn, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OHSU IRB 20645
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-01

CONDITIONS: Bleeding; Implants; Breakthrough Bleeding
Keywords: Contraceptive implant; Irregular bleeding
MeSH Terms: conditions — Hemorrhage; Metrorrhagia | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo-controlled Computer-generated randomization schema
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Placebo (oral) once daily for 30 days to be started following 3 consecutive days of bleeding
  Interventions: Drug: Placebo
- Curcumin group (Experimental): Curcumin 600 mg (oral) once daily for 30 days to be started following 3 consecutive days of bleeding
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Placebo — Placebo (oral) once daily for 30 days. Treatment to be started after 3 consecutive days of bleeding
  Arms: Placebo group
Drug: Curcumin — Curcumin 600 mg (oral) once daily for 30 days. Treatment to be started after 3 consecutive days of bleeding
  Arms: Curcumin group

SUMMARY:
The investigators plan to study the effects of curcumin, the active ingredient in the spice turmeric, on the irregular bleeding experienced by women who use the contraceptive implant.

DETAILED DESCRIPTION:
The investigators are proposing a randomized, double blind placebo-controlled clinical trial over a 30-day reference period for treatment of women experiencing bothersome bleeding while using the etonogestrel (ENG) contraceptive implant. The primary outcome of the study will be the total number of amenorrhea days in a 30-day reference period. The study has a number of secondary outcomes (see study objectives) focused around the efficacy of oral curcumin to stop bleeding/spotting and for how long.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Women 15-45 years of age
* Currently using the ENG implant for at least 30 days and use proven on exam (palpation of implant at screening visit)
* Willing to continue using the implant for at least 30 days from study enrollment
* >7 days of continuous bleeding/spotting in the last 30 days, OR 2 or more episodes of bleeding/spotting in the last 30 days.
* Access to a reliable cell phone and must be willing to receive and respond to a daily text or email message to assess bleeding and use of study drug
* Negative gonorrhea/chlamydia screening performed at screening visit

Exclusion Criteria:

* Postpartum within six months
* Post-abortion within six weeks
* Currently pregnant
* Currently breast-feeding (to be eligible, must be 4-6 weeks from cessation of breastfeeding)
* Undiagnosed abnormal uterine bleeding pre-dating placement of contraceptive implant
* Bleeding dyscrasia
* Anticoagulation use
* Active cervicitis
* Allergy to curcumin or turmeric
* History of venous thromboembolism
* Current or past breast or uterine malignancy
* Use of P450 pathway inducing drug
* Implant is due to be switched out in 2 months or less from enrollment
* Currently using oral contraceptives in addition to implant (to be eligible, needs to have a 4-6 week washout period)
* Prior pregnancy occurred while Nexplanon/Implanon was in place

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edelman A, Boniface E, Schrote K, Messerle-Forbes M, O'Donnell A, Jensen JT, Han L. Treatment of unfavorable bleeding patterns in contraceptive implant users: a randomized clinical trial of curcumin. Am J Obstet Gynecol. 2023 Aug;229(2):145.e1-145.e9. doi: 10.1016/j.ajog.2023.04.028. Epub 2023 Apr 26. PMID 37116825

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Group | Curcumin Group
Started | 29 | 29
Completed | 28 | 26
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Curcumin Group | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (3.7) | 24 (5.3) | 24 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: Asian | 3 | 1 | 4
  Race and Ethnicity: Hispanic/Latina | 2 | 8 | 10
  Race and Ethnicity: Native Hawaiian/Pacific Islander | 0 | 1 | 1
  Race and Ethnicity: White | 21 | 15 | 36
  Race and Ethnicity: More than one race | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 26 | 54
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24 (3.7) | 25 (5.1) | 24 (4.4)
Nulliparous [Count of Participants; unit: Participants] | 28 | 23 | 51

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Days Without Bleeding or Spotting
Description: Total number of days without bleeding or spotting in the 30-day reference period
Time Frame: Day 1 to Day 30
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Group | Curcumin Group
Number analyzed (Participants) | 28 | 26
days | 17.5 (4.8) | 16.7 (6.9)

2. Secondary Outcome: Total Number of Bleeding/Spotting Days
Description: Total number of days with bleeding or spotting in the 30-day reference period
Time Frame: Day 1 to Day 30
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Group | Curcumin Group
Number analyzed (Participants) | 28 | 26
days | 12.5 (4.8) | 13.3 (6.9)

3. Secondary Outcome: Total Number of Spotting Days
Description: Total number of days with spotting in the 30-day reference period
Time Frame: Day 1 to Day 30
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Group | Curcumin Group
Number analyzed (Participants) | 28 | 26
days | 4.9 (3.1) | 6.7 (4.3)

4. Secondary Outcome: Total Number of Bleeding Days
Description: Total number of days with bleeding in the 30-day reference period
Time Frame: Day 1 to Day 30
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Group | Curcumin Group
Number analyzed (Participants) | 28 | 26
days | 7.6 (4.5) | 6.6 (4.9)

5. Other Pre Specified Outcome: Change in Patient Satisfaction With Bleeding Pattern as Assessed by VAS
Description: Change in the level of patient satisfaction with bleeding pattern as measured by Visual Analog Scale (VAS) from Day 1 to Day 30. The scale ranges from 0 (lowest possible satisfaction) to 100 (highest possible satisfaction).
Time Frame: Day 1 to Day 30
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Group | Curcumin Group
Number analyzed (Participants) | 28 | 26
units on a scale | 9.5 [0.8 to 53] | 42 [18 to 64]

6. Other Pre Specified Outcome: Proportion of Participants Who Intend to Continue Use of Implant
Description: Percentage of participants who are continuing implant use or anticipate implant continuation, evaluated at the end of study
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | Curcumin Group
Number analyzed (Participants) | 28 | 26
Participants | 23 | 16

ADVERSE EVENTS:
Time Frame: Enrollment through 30 days of treatment
Arm/Group | Placebo Group | Curcumin Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 1/29 | 2/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Group (N=29) | Curcumin Group (N=29)
Stomach cramps (Gastrointestinal disorders) | 0/0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Migraine headache (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT04205929/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT04205929/ICF_001.pdf